CLINICAL TRIAL: NCT04020276
Title: A Phase I Study of OAR-Based, Dose Escalated SBRT With Real Time Adaptive MRI Guidance for Liver Metastases
Brief Title: OAR-Based, Dose Escalated SBRT With Real Time Adaptive MRI Guidance for Liver Metastases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW18110; NCI-2019-04726 (Registry Identifier: NCI Trial ID); SMPH/HUMAN ONCOLOGY/HUMAN ONCO (Other: UW Madison); A533300 (Other: UW Madison); 2019-0373 (Other: HS IRB); Protocol Version 10/28/2025 (Other: UW Madison)
Record Dates: First submitted 2019-07-11; First posted 2019-07-16 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Liver Metastases; Stereotactic Body Radiation Therapy; MRI-guided Treatment

STUDY DESIGN:
Intervention Model Description: 4+4 dose-escalation design - patients will be treated to a maximum tolerated dose using MRI-guided SBRT with real time adaptation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- MRI-Guided SBRT Dose Escalation (Experimental): Treatment on MRI Linac with SBRT in 5 fractions with adaptive planning, maximum dose 80 Gy
  Dose Escalation Bowel Pathway, V34 < 0.5cc Dose Escalation Liver Pathway, 700 cc < 16 Gy
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Participants will receive 5 fractions of radiation, which will be delivered 2-3 times per week. SBRT should be complete in a 1.5 to 2 week time frame. There should be a minimum of 12 hours between treatments.

SUMMARY:
The purpose of this trial is to identify a safe maximum tolerated dose level for MRI-guided Stereotactic Body Radiation Therapy (SBRT) treatment of bowel and liver metastases, respectively.

Eligible participants will be on study for up to 12 months.

DETAILED DESCRIPTION:
Stereotactic Body Radiation Therapy (SBRT) is a noninvasive local therapy with proven efficacy in a number of solid tumor types. The technique itself involves the precise administration of high biological equivalent dose radiation in order to maximize local control of discrete lesions.

SBRT has been shown to be an effective therapy for both primary and metastatic liver tumors of multiple histologies. In metastatic liver disease from all primary tumor sites, patients treated with modern SBRT techniques generally enjoy very high levels of 1 and 2 year local control. However, CRC liver metastases have been shown to be particularly resistant to SBRT, and often are found to have significantly worse rates of control compared with other histologies. Recent studies indicate this might be due to the inherent radioresistance of the CRC histology.

Despite this, there appears to be a relationship between increasing dose and improvement of local control, both within CRC and other tumor histologies. Higher SBRT dose was recently shown to improve local control in CRC pulmonary metastases, further corroborating the hypothesis of CRC as a radioresistant tumor. However, increasing dose delivery with SBRT has been limited based on the risk of toxicity to adjacent structures, and the ability to visualize them during treatment. This is particularly relevant in treating liver tumors, as tumor and small bowel movement can often make tumor targeting and organs-at-risk (OAR) avoidance especially difficult.

MRI-guided SBRT for liver tumors is both safe and feasible and offers an as yet unprecedented opportunity to achieve the highest possible safe dose to liver tumors.

Primary Objectives:

* To determine the safety and tolerability of using increasing bowel dose constraints for MRI-guided SBRT treatment of metastatic liver deposits from all primary histologies except as outlined in the exclusion criteria.
* To determine the safety and tolerability of using increasing volume-based liver constraints for MRI-guided SBRT treatment for metastatic liver deposits from all primary histologies except as outlined in the exclusion criteria.
* To define maximally tolerated dose constraints for both liver and bowel based on DLT using real-time, adaptive, MRI-based treatment planning.

Secondary Objectives:

* To determine local recurrence rates at 1, and 2 years using MRI-guided SBRT with dose planning from escalation of OAR constraints.
* To evaluate progression-free survival (PFS) and overall survival (OS) in this patient cohort.
* To assess quality of life and patient reported outcomes at 2 months following MRI-guided SBRT.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of histologically confirmed or clinically suspected metastatic cancer to the liver.
* Participant must be a candidate for SBRT to at least one intrahepatic lesion but no more than 6 intrahepatic lesions.
* Participant must be a candidate for treatment on the ViewRay treatment unit. Must be screened to rule out implants and devices that are not MRI compatible.
* Be willing and able to provide written informed consent.
* Participants may be therapy-naïve or have had prior systemic therapy up to two weeks prior to study entry.
* No active central nervous system (CNS) metastatic disease. NOTE: Subjects with CNS involvement must meet all of the following to be eligible:

  * At least 28 days from prior definitive treatment of their CNS disease by surgical resection, SBRT or Whole Brain Radiation Therapy (WBRT) at the time of registration
  * AND asymptomatic and off systemic corticosteroids and/or enzyme-inducing antiepileptic medications for brain metastases for >14 days prior to registration.
* Demonstrate adequate organ function as defined in the following table; all screening labs should be performed within 28 days of SBRT treatment initiation.

  * Platelet count greater than or equal to 50000 /µL
  * Absolute Neutrophil Count (ANC) greater than or equal to 1000 /µL
  * Hemoglobin (Hgb) greater than or equal to 8 g/dL or greater than or equal to 5.6 mmol/L without transfusion or erythropoietin (EPO) dependency (within 7 days of assessment)
  * Serum creatinine OR measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl) Creatinine/Calculated creatinine clearance (CrCl) greater than or equal to 30 mL/min for subject with creatinine levels greater than 1.5 X institutional upper limit of normal (ULN)
  * Bilirubin greater than or equal to 1. 5 × ULN OR direct bilirubin greater than or equal to ULN for participants with total bilirubin levels greater than 1.5 ULN
  * Aspartate aminotransferase (AST) and ALT (SGPT) greater than or equal to 5 × ULN
  * International Normalized Ratio (INR) or Prothrombin Time (PT) greater than or equal to 1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
  * Activated Partial Thromboplastin Time (aPTT) greater than or equal to 1.5 X ULN unless participant is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* For participants enrolled on the liver dose escalation arm, screening labs must be consistent with Child Pugh class A unless therapeutic anticoagulation places them in Child Pugh B. In that case, trial entry or exclusion will be at the discretion of the treating physician.
* Have a performance status of 2 or less on the Eastern Cooperative Oncology Group (ECOG) performance scale.
* Life expectancy of > 12 weeks.
* Women of childbearing potential (WOCP) should have a negative urine or serum pregnancy test prior to initiation of radiation therapy. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* WOCP must not be pregnant or breast-feeding.
* WOCP must be willing to use an effective method of birth control such as an oral, implantable, injectable, or transdermal hormonal contraceptive, an intrauterine device (IUD), use of a double barrier method (condoms, sponge, diaphragm, or vaginal ring with spermicidal jellies or cream), or total abstinence for the duration of the radiotherapy and 60 days thereafter.

NOTE: A person of childbearing potential is anyone (regardless of sexual orientation, gender identity, having undergone a tubal ligation, or remaining celibate by choice) who was born with a uterus and at least one ovary and meets both of the following criteria:

* Is post-menarcheal (i.e., has had at least one prior menses)
* Has not undergone a hysterectomy or bilateral oophorectomy or has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Participant is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the initiation of SBRT.
* History of a second invasive cancer in the last 3 years (except for appropriately treated low-risk prostate cancer, treated non-melanoma skin cancer, appropriately treated ductal carcinoma in situ or early stage invasive carcinoma of breast appropriately treated in situ/early stage cervical/endometrial cancer.
* Has an active infection requiring systemic therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with follow up scans or visits.
* Has a primary tumor histology of germ cell tumor, leukemia, or lymphoma.
* Has a primary liver cancer such as cholangiocarcinoma or hepatocellular carcinoma.
* Has had prior radiation therapy that significantly overlaps with the liver.
* Has a diagnosis of Crohn's disease, ulcerative colitis, or scleroderma.
* Participants with Gilbert's disease or other primary disorders of bilirubin metabolism will not be allowed on the trial.
* For participants in the liver dose escalation arm only, has pre-existing liver disease such that patients are classified as Child Pugh B or worse. If the participant is anti-coagulated such that their INR places them in the CP-B classification, exclusion or inclusion will be at the discretion of the treating physician.
* Pregnancy or women of childbearing potential and men who are sexually active and refuse to use medically acceptable forms of contraception.
* Participants with implanted hardware that would preclude MRIs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2019-11-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Acute Dose Limiting Toxicity (DLT) | Up to 4 weeks
  Dose limiting toxicity (DLT) will be defined as grade 3 or greater* non-hematologic toxicity attributable to radiation therapy, and occurring within 4 weeks after the completion of SBRT.
  *With the exception of liver function tests, which are allowed up to and including grade 3

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 5 years
  Progression-free survival (PFS) will be defined as the difference (in months) between the date of study enrollment and the date of disease progression or death due to any cause
Overall Survival (OS) | Up to 5 years
  Overall survival (OS) will be defined as the difference (in months) between the date of study enrollment to the date death due to any cause.
Local Control Rates | up to 2 years
  Point estimates along with the exact 95% confidence interval will be computed for the local control rates
Change in Quality of Life (QoL) | Baseline, 2 months (1 month post treatment follow-up)
  QoL will be assessed on a 5 item questionnaire using a 4-point Likert scale, where 4 = Not at all and 1 = Constant. Scores range from 5-20 where higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bassetti, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu